CLINICAL TRIAL: NCT00584649
Title: Ablation of Inappropriate Sinus Tachycardia Syndrome by Targeting Cardiac Neural Input
Brief Title: Ablation of Inappropriate Sinus Tachycardia
Acronym: IST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed out when PI left the university.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1364
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Inappropriate Sinus Tachycardia
Keywords: Inappropriate Sinus Tachycardia; Inappropriate Tachycardia; Sinus Tachycardia; Palpitations; Fast Heart rate
MeSH Terms: conditions — Tachycardia, Sinus; Tachycardia | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Other): electrophysiology study and radiofrequency ablation
  Interventions: Procedure: electrophysiology study and radiofrequency ablation

INTERVENTIONS:
Procedure: electrophysiology study and radiofrequency ablation — stimulation protocol searching for the neural inputs to the sinus node region and radiofrequency ablation of neural input to the heart

SUMMARY:
Hypothesis- Radiofrequency ablation, targeting the sympathetic input of the sinus node identified by 20Hz stimulation at the junction of the superior vena cava and the right atrium, will effectively reduce sinus rate acutely and will reduce palpitations due to inappropriate sinus tachycardia without the need for pacemaker implantation due to sinus node dysfunction post ablation.

DETAILED DESCRIPTION:
Inappropriate sinus tachycardia syndrome describes a condition in which a patient's heart rate is intermittently (or persistently) higher than expected for the physiological circumstances, with ECG appearance indistinguishable from normal sinus rhythm, after the exclusion of medical conditions causing sinus tachycardia.

Hypothesis- Radiofrequency ablation, targeting the sympathetic input of the sinus node identified by 20Hz stimulation at the junction of the superior vena cava and the right atrium, will effectively reduce sinus rate acutely and will reduce palpitations due to inappropriate sinus tachycardia without the need for pacemaker implantation due to sinus node dysfunction post ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 80 years old, who are scheduled for an ablation procedure for suspected inappropriate sinus tachycardia, with symptomatic palpitations during periods where documented electrogram recordings suggest sinus tachycardia (holter, event recorder, or 12 lead ECG).
2. Sinus rate greater than 100 bpm with minimal physiologic challenge, or mean sinus rate during 24 hour holter more than 95bpm, or daytime resting heart rate more than 95bpm.
3. Symptoms (or sinus rate) not explained by an alternative medical or electrophysiological diagnosis.
4. Symptoms refractory to treatment with beta-blocker medication, or beta-blockers contra-indicated or not tolerated

Exclusion Criteria:

1. Children under 18 years of age (due to greater risk from exposure to X rays).
2. Any medical condition significantly increasing the risk of extending the ablation procedure or of X ray exposure, including pregnancy.
3. Significant orthostatic hypotension (due to need for rapid chronotropic response to fall in blood pressure)
4. An alternative cause for sinus tachycardia identified (e.g. hyperthyroidism or pheochromocytoma).
5. Inability or unwillingness to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Improvement in:symptoms(palpitations);quality of life;resting heart rate;mean 24 hour heart rate;heart rate variability; | Clinical efficacy is established if the improvement is maintained after 6months to a year.

SECONDARY OUTCOMES:
duration of symptom limited Bruce protocol exercise treadmill test;duration of exercise test required to increase rate by 20%. | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Lockwood, MD, Principal Investigator — University of Oklahoma HSC Assistant Professor Medicine/Cardiology
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States